CLINICAL TRIAL: NCT06441864
Title: Behavioral Treatment for Nightmares in REM Sleep Behavior Disorder
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 00187090; 09-SRG-23 (Other Grant/Funding Number: Sleep Research Society Foundation)
Record Dates: First submitted 2024-05-28; First posted 2024-06-04 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: Nightmare; Nightmare Disorder With Associated Other Sleep Disorder; REM Sleep Behavior Disorder
Keywords: Imagery Rehearsal Therapy; Cognitive Behavioral Therapy for Nightmares
MeSH Terms: conditions — REM Sleep Behavior Disorder | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Intervention Model Description: Multiple baseline single case experimental design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 2-week baseline (Experimental): Participants will receive treatment after a 2-week baseline assessment period
  Interventions: Behavioral: Cognitive Behavioral Therapy for Nightmares
- 4-week baseline (Experimental): Participants will receive treatment after a 4-week baseline assessment period
  Interventions: Behavioral: Cognitive Behavioral Therapy for Nightmares

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy for Nightmares — The intervention will consist of 7 therapy sessions (once per week for 7 weeks) which will be delivered via videoconference. Partners will attend 2 of the 7 treatment sessions. During the sessions, participants will learn techniques for managing and changing nightmares.
  Other Names: Imagery Rehearsal Therapy

SUMMARY:
The purpose of this clinical trial is learn whether a behavioral (non-medication) treatment can reduce nightmares in adults with Rapid Eye Movement (REM) Sleep Behavior Disorder (RBD). People with RBD will be enrolled in the study along with their romantic partners. All participants will receive the treatment via videoconference and will complete 2 assessments. Participants with RBD will attend 7 sessions, and their partners will attend 2 of those sessions with them.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of isolated RBD or RBD secondary to neurodegenerative disease
* Age 18 or older
* Speak, read, and write English
* Live in the United States
* Nightmare frequency ≥3 times per week
* Disturbing Dream and Nightmare Severity Index score indicative of nightmare disorder
* Sleep, neurological, and psychiatric medications stable for at least 1 month and willing to keep medications stable through the course of the study
* Live with a romantic partner who is willing to participate in the study

Exclusion Criteria:

* Possible dementia
* Narcolepsy
* Posttraumatic stress disorder
* Previous behavioral treatment for nightmares
* Currently engaged in sleep- or trauma-focused psychotherapy
* Taking a medication that could cause RBD, if the medication was started prior to onset of RBD symptoms

Inclusion Criteria (Partners):

* Live with a romantic partner who meets all of the above criteria
* Age 18 or older
* Speak, read, and write English
* Live in the United States

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-07-15 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Disturbing Dream and Nightmare Severity Index (DDNSI) | Baseline and posttreatment
  The DDNSI is a questionnaire which measures the severity of nightmares.
Nightmare frequency (sleep diary) | Baseline and posttreatment
  The number of nightmares experienced each day will be collected on daily sleep diaries completed during each assessment period.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Utah, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No